CLINICAL TRIAL: NCT05978752
Title: Clinical Study on Endoscopic Management of GOV1 Esophagogastric Varices Based on CT Hemodynamics
Brief Title: Clinical Study on Endoscopic Management of GOV1 Esophagogastric Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jinhua Hospital Affiliated to Zhejiang University (Unknown); Lanxi People's Hospital (Other); Lishui Country People's Hospital (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0437
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-07

CONDITIONS: Esophageal and Gastric Varices
Keywords: GOV1 esophagogastric varices; HVPG; endoscopic treatment
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Intervention Model Description: The patients with GOV1 esophagogastric varices were treated with gastric variceal tissue gel injection, at the same time, the esophageal varices were treated with ligation, sclerotherapy, or no treatment. A new method for the treatment of esophageal varices was proposed to improve the effective rate and reduce the recurrence rates and mortality, shorter hospital stays, and lower treatment costs, while further expanding the value of HVPG testing.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Active Comparator): The patients will undergo endoscopic gel embolization of gastric fundus varices and esophageal varices ligation.
  Interventions: Procedure: Endoscopic gel embolization of gastric fundus varices and ligation of esophageal varices
- B (Active Comparator): The patients will undergo endoscopic gel embolization of gastric fundus varices and sclerotherapy of esophageal varices.
  Interventions: Procedure: Endoscopic gel embolization of gastric fundus varices and sclerotherapy of esophageal varices
- C (Experimental): The patients will undergo endoscopic gelatinization of gastric varices (esophageal varices were not treated).
  Interventions: Procedure: Endoscopic gelatinous embolization of gastric varices (esophageal varices not treated)

INTERVENTIONS:
Procedure: Endoscopic gel embolization of gastric fundus varices and ligation of esophageal varices — For patients with GOV1 esophagogastric varices, gastric varices will be treated with endoscopic gelatinous embolization, esophageal varices will be treated with ligation.
  Arms: A
Procedure: Endoscopic gel embolization of gastric fundus varices and sclerotherapy of esophageal varices — For patients with GOV1 esophagogastric varices, gastric varices will be treated with endoscopic gelatinous embolization, esophageal varices will be treated with sclerotherapy.
  Arms: B
Procedure: Endoscopic gelatinous embolization of gastric varices (esophageal varices not treated) — For patients with GOV1 esophagogastric varices, only gastric varices will be treated with endoscopic gelatinous embolization, esophageal varices will not be treated.
  Arms: C

SUMMARY:
The patients with GOV1 esophagogastric varices will be treated with gastric variceal tissue gel injection, at the same time, the esophageal varices were treated with ligation, sclerotherapy, or no treatment. A new method for the treatment of esophageal varices will be proposed to improve the effective rate and reduce the recurrence rates and mortality, shorter hospital stays, and lower treatment costs, while further expanding HVPG testing to develop the best strategy for secondary prevention of endoscopic treatment in patients with GOV1 type esophageal and gastric varices.

DETAILED DESCRIPTION:
Cirrhotic portal hypertension can cause esophageal and gastric varices, and esophageal and gastric varices bleeding (EGVB) were associated with portal vein pressure. At present, the gold standard for detecting portal pressure in clinical practice is hepatic venous pressure gradient (HVPG). For Sarin classification GOV1 of esophagogastric varices are from a single origin, the left gastric vein. If the fundus varicose veins receive complete embolization treatment, the esophageal variceal blood flow should be completely blocked, and such patients do not need to perform esophageal surgery. However, this has not been reported in the literature.

Patients with esophageal and gastric varices identified by CT as GOV1 will be enrolled, all of whom will receive HVPG detects. The patients were randomly divided into three groups. The patients in group A will receive endoscopic gel embolization for gastric varices and esophageal varices ligation treatment, group B patients will receive endoscopic gastric variceal tissue glue embolization and esophageal variceal sclerotherapy treatment, the patients in group C will receive endoscopic gelatinization of gastric fundus varices (esophageal varices were not treated). Patients in the three groups were followed up with CTP and gastroscopy 1 month, 3 months, and 6 months after the initial treatment, and additional endoscopic treatment will be provided if necessary. If bleeding occurs again during this period, timely treatment (medication, endoscopy, intervention or surgery) is required according to the condition.

A new method for the treatment of esophageal varices will be proposed to improve the effective rate and reduce the recurrence rates and mortality, shorter hospital stays, and lower treatment costs, while further expanding HVPG testing to develop the best strategy for secondary prevention of endoscopic treatment in patients with GOV1 type esophageal and gastric varices.

ELIGIBILITY:
Inclusion Criteria:

* GOV1 esophageal and gastric varices identified by CT; more than 18 years old;

Exclusion Criteria:

* Complicated with liver cancer, severe cardiopulmonary insufficiency, stage III and above hepatic encephalopathy, severe natural portal shunt formation, and previous treatment of portal hypertensive bleeding (including endoscopic, interventional, and surgical procedures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
hemostasis rate | 6 month
  the percentage of hemostasis

SECONDARY OUTCOMES:
Postoperative bleeding recurrence rate | 6 month
  Rebleeding rate after endoscopic treatment: including hematemesis and/or black stool, hemoglobin decrease >10g/L

CONTACTS AND LOCATIONS:
Overall Officials: Wei Li, Master, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Liangjing Wang, Doctor, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China